CLINICAL TRIAL: NCT05034991
Title: The Role of Endometrial Blood Flow in Endometrial Cancer
Status: Recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 109171-E
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of endometrial cancer is gradually increasing nowaday. Sonography can be used to evaluate the endometrial volume, the vascularity and the blood flow. This study will analyze the role of preoperative endometrial blood flow in the outcome of endometrial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

- >20 years old female had Endometrial cancer

Exclusion Criteria:

- <20 years old female

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: endometrial cancer patient
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between the endometrial vascularity (VFI, FI, VI), endometrial volume, endometrial thickness and progression-free survival of endometrial cancer patients | 12 months
  Correlation between the endometrial vascularity (VFI, FI, VI), endometrial volume, endometrial thickness and progression-free survival of endometrial cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan